CLINICAL TRIAL: NCT05299814
Title: The Impact of Parental Emotion Regulation Capacity on Behavioral Treatment for Pediatric ADHD
Brief Title: Impact of Parental Emotion Regulation on the Treatment of ADHD
Acronym: PERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, James Waxmonsky, Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERS
Record Dates: First submitted 2022-02-10; First posted 2022-03-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: ADHD
Keywords: oppositional behaviors, conduct problems
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: single group open label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavior Therapy (Experimental): 8 sessions of an evidence based parenting program to address oppositional behaviors and ADHD symptoms at home. All participants are in this arm.
  Interventions: Behavioral: Behavioral Parenting Intervention

INTERVENTIONS:
Behavioral: Behavioral Parenting Intervention — 8 session evidence based parenting intervention

SUMMARY:
Aim: To examine if parental emotion regulation (ER) moderates the response to parent training interventions.

H1: Reduced parental ER capacity will predict diminished efficacy for behavioral parent training to improve negative parenting behavior (NPB) and behavior problems in offspring with ADHD.

H2: Increased parental emotional reactivity will predict diminished efficacy for behavioral parent training to improve negative parenting behavior (NPB) and behavior problems in offspring with ADHD.

DETAILED DESCRIPTION:
Children ages 5-12 with ADHD and at least a mild level of oppositional behaviors will be enrolled in a single arm study examining the impact of objective and self rated measurements of parental emotion regulation and emotional reactivity to predict the degree of improvement seen in children's oppositional behaviors and negative parenting behaviors and from an evidence based eight session parenting intervention. The program emphasizes attending to positive behavior, contingent rewards for good behaviors and predictable consequences, such as time-out or loss of privilege, for negative behaviors. The primary outcome is change in parent ratings of symptoms of Oppositional Defiant Disorder (ODD) as measured by the Disruptive Behaviors Disorder Rating Scale (DBDRS).Negative parenting behaviors (NPB) will be assessed using the Alabama Parenting Questionnaire which measures five different domains of parenting and has been used in past trials to detect changes in NPB. Measures will be collected at baseline, midpoint and endpoint. Parental ER capacity will be examined as moderators of the treatment effect on children's symptom levels and NPB.

We will employ two measures of parental emotion regulation: self report using the Difficulties with Emotion Regulation Scale (DERS) and the change in amplitude on the late positive potential (LPP) during an emotion regulation task. The total score from the DERS collected at baseline will serve as the self report measure of parental ER. The total score is the sum of the 6 DERS subscales: nonacceptance of emotional responses, difficulties engaging in goal directed behavior, impulse control difficulties, lack of emotional awareness, limited emotion regulation strategies and lack of emotional clarity.

A cognitive reappraisal task completed under EEG monitoring will serve as the neurobiological measurement of emotion regulation capacity. Change in LPP amplitude on this task has been well established as measure of regulatory capacity. The stimulus set will be comprised of 30 unpleasant, high arousing and 30 neutral, low arousing images from the International Affective Picture System (IAPS). The study will consist of 1 block of 90 stimuli with three types of randomly ordered trials within the block. There will be 30 trials each of a "look neutral", "look negative" and "decrease negative" trial (described below). On each trial, participants will first be asked to relax (baseline) prior to seeing a cue word for 2 seconds on the screen telling them either to "look" or "decrease." After the cue word, a fixation cross to orient visual attention is shown for 500ms, followed by the stimulus for 6 seconds. After each picture, participants will rate their level of arousal on a 0-7 likert. There will be a 2.5 second pause between trials. Prior to data collection, there will be two practice blocks. In the first, participants are given explicit instructions on what to do during the look and decrease trials, with examples of appropriate reappraisal. For 5 practice trials, they will be given detailed feedback on their appraisal efforts. The second practice will consist of 10 trials mimicking the exact procedures for the real task (no feedback). Emotion regulation capacity will be defined as the change in the LPP amplitude between the "look negative" and "decrease negative" trials, with "look neutral" vs look negative" serving as reference comparison to measure the participants' reactivity to emotional stimuli. Total task time is estimated to be 20-22 minutes. On the "decrease negative" trials, participants will be advised to create a positive frame for the story in order to feel negative emotions less strongly. For example, if shown a picture of a corpse, one could imagine that a crime had been solved preventing future murders. In the "look negative" trials, participants will be advised not to perform any reappraisal and simply rate the picture as they see it. In all trials, participants will be instructed only to think about the picture and not to intentionally distract themselves.

Electroencephalogram (EEG) data will be recorded using a 32-channel BrainProducts actiCHamp system and BrainVision Recorder software with electrodes placed over the left and right mastoids as reference electrodes, and above and below the eyes to measure the electrooculogram. The EEG signal will be digitized at 24-bit resolution and sampled at 500 Hz. Data will be processed using BrainVision Analyzer software, and segmented 200ms prior to stimulus onset and continuing for the 6 sec stimulus duration. Data will be referenced to the mastoid averages, filtered from .01 to 30 Hz, and corrected for artifacts. Event-related brain potentials (ERPs) will be constructed by separately averaging "look neutral", "look negative" and "decrease negative" trials for each recording site. The average activity in the 200ms window prior to cue onset will be the baseline. LPP amplitude will be defined as the average amplitude at central-parietal electrodes where LPP is maximal. Consistent with prior work and to evaluate changes in LPP across time as a function of reappraisal, LPP will be examined in in frontal and parietal sites at early (400 to 700ms after image onset), middle (700 to 1000ms) and late (1000 to 6000ms) time windows. Mean LPP amplitudes will be exported from BrainVision and evaluated with SPSS.

After completing this task, participants will also complete the Emotional Faces Task while undergoing EEG assessment using the same EEG techniques and ERP outcomes described above to measure the neurophysiological response to emotions (emotional reactivity). During the task, participants will view images of children with angry or neutral emotional expressions from the NIMH child faces stimulus set or pixelated faces in which the expression is unclear. Following the emotional face, an arrow (< or >) briefly appears on the screen and participants are instructed to press a mouse button to correspond with the direction of the arrows in order to ensure participants are attending to the images. Finally, the same emotional face is presented briefly so that the arrow appears between presentations of the same stimulus. Participants will first complete a brief practice block and then will view complete the emotional faces task. Consistent with prior work measuring reactivity to facial stimuli, LPP change between angry and pixleated faces will be examined in in occipital and parietal sites between 300 to 1000ms after image onset.

This study will examine if parental emotion regulation capacity is associated with the degree of symptomatic improvement in children's oppositional behaviors and negative parenting behaviors (NPB) following a course of behavioral parent training, and whether this association is moderated by parent emotional regulation or parent emotional reactivity. It is hypothesized the association between negative parenting behaviors will be more strongly associated with negative child behavior for parents with lower capacities for emotion regulation (as measured by smaller changes in LPP amplitude/higher scores on the DERS). This hypothesis will be tested by computing multilevel model, with treatment (pre, post) as the level 1 (within-subjects) predictor and parent ER as the level-2 (between-subjects) predictors, along with parent and child demographics as covariates. Separate analyses will be conducted for child and parent outcomes. Analyses will then be repeated using the objective measure of parental emotional reactivity (LPP amplitude change during the faces task) as the moderator in place of parental emotional regulation capacity.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child ages 5-12 with ADHD
* Parent must report that the child has at least a mild level of symptoms at home of Oppositional Defiant Disorder (ODD) on the Disruptive Behavior Disorder Rating Scale (DBDRS)

Exclusion Criteria:

1. Not being the parent of a child ages 5-12 who meets diagnostic criteria for ADHD.
2. Non English Speaking
3. the child with ADHD has a diagnosis of intellectual delay or has prominent autistic traits
4. Another child in the same family participating in this study already
5. Parent does not have a smartphone or tablet device to complete EMA ratings or does not reside with child for the majority of the time.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2017-04-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oppositional Defiant Disorder Symptoms (change from baseline to endpoint) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent ratings of symptoms of Oppositional Defiant Disorder as rated on the Disruptive Behavior Disorder Rating Scale (DBD-RS). The Oppositional Behavior subscale on the DBD-RS measures 8 items rated 0-3. Items are averaged to create a mean total score between 0-3. Higher scores indicate greater impairment and worse outcomes.

SECONDARY OUTCOMES:
Change in ADHD symptoms (change from baseline to endpoint) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent ratings of symptoms of ADHD as rated on the Disruptive Behavior Disorder Rating Scale. The ADHD symptom subscale on the DBD-RS has 18 items rated 0-3 that are averaged to create a mean total score (0-3). Higher scores indicate greater impairment and worse outcomes.
Change in Conduct Disorder Symptoms (change from baseline to endpoint) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent ratings of symptoms of Conduct Disorder as rated on the Disruptive Behavior Disorder Rating Scale (DBD-RS). The Conduct Disorder subscale on the DBD-RS conduct scale has 15 items rated 0-3 that are averaged to create a mean total score (0-3). Higher scores indicate greater impairment and worse outcomes.
Change in Irritability symptoms (change from baseline to endpoint) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent ratings of symptoms of irritability as rated on the Disruptive Behavior Disorder Rating Scale (DBD-RS). The Irritability symptom subscale on the DBD-RS has 3 items rated 0-3. They are averaged to create a mean total symptom score (0-3). Higher scores indicate greater impairment and worse outcomes.
Change in rates of Poor Monitoring from Baseline (before therapy) to Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent self-report ratings of poor monitoring as rated on the Alabama Parenting Questionnaire (APQ). The Poor Monitoring subscale on the APQ has 10 items rated 1-5. They are summed to create a total score. Higher scores indicate greater impairment and worse outcomes.
Change from Baseline (before therapy) Inconsistent Discipline at Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent self-report ratings of inconsistent discipline as rated on the Alabama Parenting Questionnaire (APQ). The Inconsistent Discipline subscale on the APQ has 6 items rated 1-5. Scores from each item are summed to create a total score. Higher scores indicate greater impairment and worse outcomes.
Change from Baseline (before therapy) Corporal Punishment at Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent self-report ratings of corporal punishment as rated on the Alabama Parenting Questionnaire (APQ). This subscale on the APQ has 3 items rated 1-5. Scores from each item are summed to create a total score. Higher scores indicate greater impairment and worse outcomes.
Change from Baseline (before therapy) Parental Involvement at Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent self-report ratings of parental involvement as rated on the Alabama Parenting Questionnaire (APQ). The Poor Monitoring subscale on the APQ has 10 items rated 1-5. Scores from each item are summed to create a total score. Higher scores indicate greater impairment and worse outcomes.
Change from Baseline (before therapy) Positive Parenting at Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent self-report ratings of positive parenting as rated on the Alabama Parenting Questionnaire (APQ). This subscale on the APQ has 6 items rated 1-5. Scores from each item are summed to create a total score. Higher scores indicate greater impairment and worse outcomes.
Change from Baseline (before therapy) Overall Impairment at Endpoint (after last therapy session) | baseline (week 0 prior to first therapy session), endpoint (after 8th therapy session which on average is 12 weeks later ))
  This will be measured using parent ratings of overall impairment as rated on the Impairment Rating Scale (IRS). The Overall Impairment subscale on the IRS has a minimum score of 0 and maximum score of 6. Higher scores indicate greater impairment and worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Dept of Psychiatry, Hershey, Pennsylvania, United States